CLINICAL TRIAL: NCT05532501
Title: Differential Modulation of Neural and Behavioral Responses to Emotional Scenes by Intranasal and Oral Oxytocin Administration in Healthy Men
Brief Title: The Effects of Intranasal and Oral Administration of Oxytocin on Responses to Emotional Scenes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-91
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Oral; Intranasal; Oxytocin; Emotional processing
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind between-subject design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral Oxytocin (Active Comparator): Administer oxytocin (24 IU) orally
  Interventions: Drug: Oral Oxytocin
- Intranasal Oxytocin (Active Comparator): Administer oxytocin (24 IU) intranasally
  Interventions: Drug: Intranasal Oxytocin
- Oral placebo (Placebo Comparator): Administer placebo orally (identical ingredients, except the active agent)
  Interventions: Drug: Oral placebo
- Intranasal placebo (Placebo Comparator): Administer placebo intranasally (identical ingredients, except the active agent)
  Interventions: Drug: Intranasal placebo

INTERVENTIONS:
Drug: Oral Oxytocin — Administer oxytocin (24 IU) orally, 6 individual 0.1 ml puffs (4 IU/0.1ml) on the tongue (lingual), one every 30 seconds
  Other Names: Oxytocin orally
  Arms: Oral Oxytocin
Drug: Intranasal Oxytocin — Administer oxytocin (24 IU) intranasally, 6 individual 0.1 ml puffs (4 IU/0.1ml), three puffs per nostril one every 30 seconds
  Other Names: Oxytocin intranasally
  Arms: Intranasal Oxytocin
Drug: Oral placebo — Administer placebo orally, 6 individual 0.1 ml puffs on the tongue (lingual), one every 30 seconds.
  Other Names: Placebo orally
  Arms: Oral placebo
Drug: Intranasal placebo — Administer placebo intranasally, 6 individual 0.1 ml puffs, three puffs per nostril one every 30 seconds
  Other Names: Placebo intranasally
  Arms: Intranasal placebo

SUMMARY:
The study will investigate whether oxytocin administered either intranasally or orally (lingual) (24 international units, IU) can differentially modulate men's neural and behavioral responses to emotional scenes using an implicit emotional paradigm.

DETAILED DESCRIPTION:
Previous studies have reported that oxytocin administration intranasally and orally (spray on the tongue) can modulate neural and behavioral responses during processing of face emotions and can influence top-down attention to social stimuli. However, no research has directly compared the neural and behavioral effects of the two different administration routes on the processing of emotional scenes. In the current randomized, double-blind, between-subjects, placebo-controlled study, 160 healthy male subjects will be recruited and receive treatment either oxytocin (24IU, orally/intranasally) or placebo (orally/intranasally). Prior to treatment, all subjects will complete a number of questionnaires to control for potential group differences in potential confounders in terms of personality traits and mood, including: Beck Depression Inventory-II (BDI), Autism Spectrum Quotient (ASQ), Liebowitz Social Anxiety Scale (LSAS), State-Trait Anxiety Inventory (STAI), Childhood Trauma Questionnaire (CTQ), Interpersonal Reactivity Index (IRI). Additionally, the Positive and Negative Affect Schedule (PANAS) is administered before the treatment and before and after completing the implicit emotional scanning task to measure any changes in mood. Forty-five minutes after receiving treatment, subjects will be required to undergo and MRI scanning session including structural scans and resting-state fMRI followed by an implicit emotional scene processing task (picture source: Nencki affective picture system, including positive, neutral, and negative-valence social and non-social scenes). After fMRI scanning, subjects will be required to rate emotional stimuli presented during the scan on valence, intensity, and arousal using 1-9 point Self-Assessment Manikin (SAM) scales.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

* 1. History of brain injury 2. Head trauma 3. Substance abuse 4. Medication

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Compare the effects of oxytocin on neural responses to emotional scenes between intranasal and oral administration routes. | 45~70 minutes after treatment
  Comparison of whole brain neural (fMRI scanning) activation differences between oral and intranasal oxytocin administration to emotional scenes will be performed using a mixed ANOVA with route (oral/intranasal), treatment (oxytocin/placebo) as between subject factors and valence of emotional scenes (positive/negative/neutral) as within-subject factor, post-hoc comparisons will be conducted to further disentangle the significant interactions observed after the mixed ANOVA.
Compare the effects of oxytocin on behavioral responses to emotional scenes between intranasal and oral administration routes. | 70~90 minutes after treatment
  Differences in behavioral ratings of valence (1-9 point Self-Assessmen-Manikin (SAM) scale, 1 means very negative, 9 means very positive, 5 means neutral), intensity (1-9 point SAM scale, 1 means mild, 9 means strong), and arousal (1-9 point SAM scale, 1 means not aroused at all, 9 means very aroused) of emotional scene stimuli between oral oxytocin and intranasal oxytocin groups will be examined using mixed ANOVAs, respectively.

SECONDARY OUTCOMES:
Compare the effect of oxytocin on neural functional connectivity during processing of emotional scenes between intranasal and oral administration routes. | 45~70 minutes after treatment
  Comparison of functional connectivity (fMRI scanning) differences between oral and intranasal oxytocin administration to emotional scenes by means of a mixed ANOVA with route (oral/intranasal), treatment (oxytocin/placebo) as between subject factors and emotional scene (positive/negative/neutral) as within-subject factor, post-hoc comparisons was conducted to further disentangle the significant interaction observed after mixed ANOVA.
Correlations between neural activation and behavioral effects of intranasal or oral oxytocin during emotional scene processing. | 45~90 minutes after treatment
  Pearson correlation tests will be used to compute correlations between any significant neural and behavioral effects of treatment.
Correlations between functional connectivity and behavioral effects of intranasal or oral oxytocin during emotional scene processing. | 45~90 minutes after treatment
  Pearson correlation tests will be used to compute correlations between any significant neural and behavioral effects of treatment.
Comparison of effects of oxytocin on pre-task resting-state functional connectivity (rsfMRI) between intranasal and oral administration routes. | 45~70 minutes after treatment
  Comparisons of whole brain rsfMRI will be performed using an ANOVA with route (oral/intranasal) and treatment (oxytocin/placebo) as between-subject factors. Post-hoc comparisons will be used to disentangle significant interactions observed in the ANOVA.
Mood changes assessed by the Positive Affect Negative Affect Schedule (PANAS) in all treatment groups during the experiment. | 0~70 minutes
  The Positive Affect Negative Affect Schedule measures both positive and negative mood in a person. The Positive Affect score ranges from 10-50, with higher scores representing higher levels of positive affect. The Negative Affect scores range from 10-50, with lower scores representing lower levels of negative affect. The differences in PANAS scores at each time-point between treatment groups will be analyzed using mixed ANOVAs.

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- school of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China